CLINICAL TRIAL: NCT00587860
Title: A Placebo-Controlled Trial of St. John's Wort for Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Yuri A. Saito Loftus, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 132-06
Record Dates: First submitted 2007-12-27; First posted 2008-01-08 (Estimated); Results first posted 2010-03-01 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Hypericum extract LI 160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- St. John's Wort (Active Comparator)
  Interventions: Drug: St. John's wort

INTERVENTIONS:
Drug: St. John's wort — Dosage form: Tablet (450 mg) Dose: 450 mg twice a day, placebo twice a day
  Other Names: Latin name: Hypericum perforatum L.; Common name: St. John's Wort
  Arms: St. John's Wort
Drug: Placebo — Dosage form: Tablet (450 mg) Dose: 450 mg twice a day, placebo twice a day
  Arms: Placebo

SUMMARY:
This study is being done to see if St. John's wort helps people with irritable bowel syndrome, otherwise known as "IBS". St. John's wort is a herbal supplement derived from the St. John's wort plant. It has been shown to be helpful in several medical conditions such as depression as well as other pain syndromes.

DETAILED DESCRIPTION:
Eligibility criteria:

1. Established diagnosis of IBS
2. 18-70 years of age

4) U.S. resident 5) English-speaking (able to provide consent and complete questionnaires) 6) Able to participate in all aspects of the study

You will be asked to do the following:

* Undergo a screening interview and physical examination
* Take a urine pregnancy test (if applicable)
* Take a study pill twice daily for 12 weeks(3 months)
* Complete daily symptom diaries and bi-weekly questionnaires for 12 weeks.
* Complete a questionnaire at 6 months after the active phase of the study is over.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of IBS
* Meet Rome II diagnostic criteria for IBS
* 18-70 years of age
* U.S. resident
* English-speaking (able to provide consent and complete questionnaires)
* Able to participate in all aspects of the study

Exclusion Criteria:

* Known alternative/concurrent gastrointestinal diagnosis (e.g. Crohn's disease, ulcerative colitis, microscopic colitis, celiac sprue, chronic pancreatitis or pancreatic insufficiency, scleroderma, chronic intestinal pseudo-obstruction, bacterial overgrowth, recent (<6 months) intestinal bacterial/protozoal/ parasitic infections, HIV, fecal incontinence, small bowel or colonic resection, pelvic floor dysfunction, paraplegia or quadriplegia)
* Current symptoms of severe depression, as measured by Center for Epidemiological Studies Depression Scale (CES-D) score
* Mental retardation or any condition requiring a legal guardian
* Current or past history of psychotic disorder (schizophrenia, bipolar disorder)
* Recent or current use (within past 30 days) of select mood or pain or symptom-altering medications:

  * benzodiazepine use
  * substance abuse
  * narcotic use
  * antihistamine use
  * barbiturates
  * zaleplon (Sonata)
* Recent or current use (within past 30 days) of drugs that interact with SJW:

  * antidepressants or antipsychotics
  * tramadol (Ultram)
  * sumatriptan (Imitrex)
  * digoxin (Lanoxin)
  * anticonvulsants (e.g. carbamazepine or phenytoin)
  * immunosuppressants: cyclosporine and tacrolimus
  * HIV protease inhibitors (e.g. indinavir), non-nucleoside reverse transcriptase inhibitors (e.g. nevirapine)
  * warfarin (Coumadin)
  * theophylline
  * chemotherapy
  * sulfa-containing drugs
  * piroxicam (Feldene)
  * simvastatin (Zocor)
  * sibutramine (Meridia)
  * verapamil (Calan or Isoptin)
* Planned surgery (especially transplant) or anesthesia exposure during trial
* Known photosensitivity or planned photodiagnostic or phototherapy procedures
* Are pregnant, lactating, likely to become pregnant during medication phase and not willing to use a reliable form of contraception (barrier contraceptives, diaphragm, injections, intrauterine device, surgical sterilization, and abstinence)
* Recent or current use (within 30 days) of SJW, other herbal products for IBS, investigational drug use
* Known allergy to SJW
* Significant acute or chronic progressive neurologic, hepatic, renal, cardiovascular, respiratory or metabolic disease
* Recent history of alcohol or substance dependence use or abuse
* Another household member or relative participating in the study
* Professional drivers or operators of heavy machinery
* Major cardiovascular events in the last 6 months
* Use of IBS-specific drugs such as tegaserod (Zelnorm) and Lotronex (Alosetron) (within 30 days)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri A. Saito Loftus, M.D. M.P.H., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified through community, institutional advertisement, clinicaltrials.gov, through the IFFGD webpage as well as through the outpatient clinics beginning in February 2006. Participants who participated in previous IBS studies were also mailed a recruitment letter to ask if they would be interested in participating.
Pre-assignment Details: For this study, there was a 2-week screening and enrollment phase. During this period, participants were screened, a symptom questionnaire was completed, and there was a physician exam. After the in-person screening visit, a phone call was made prior to mailing the study materials to ensure the participant was still willing to participate.
Groups:
- St. John's Wort: St. John's Wort, 450 mg twice a day
- Placebo: Placebo, twice a day
Period: Overall Study
Arm/Group | St. John's Wort | Placebo
Started | 35 | 35
Completed | 30 | 30
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | St. John's Wort | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 35 | 68
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 42.2 (14.34) | 39.43 (11.26) | 40.81 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
Bowel Symptom Score (BSS) [Median (Full Range); unit: Units on a scale] — The BSS is a five question, 100-mm visual analog scale of four IBS symptoms (pain/discomfort, bloating, constipation, and diarrhea), and an overall severity scale. The best possible value would be 0 (no symptoms) and the worst is 500 (severe symptoms). BSS was assessed on a bi-weekly basis.
  Units on a scale | 173 [36 to 314] | 165 [73 to 290] | 169 [36 to 314]
Center for Epidemiologic Studies Depression Scale (CES-D) score [Median (Full Range); unit: Units on a scale] — We measured CES-D Score at baseline as well as bi-weekly throughout the study. The CES-D is a self-reported 20 question survey designed to measure depressive symptomatology in the general population. The possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
  Units on a scale | 6 [0 to 26] | 5 [0 to 32] | 5.5 [0 to 32]
Irritable Bowel Syndrome - Quality of Life (IBS-QoL) [Median (Full Range); unit: Units on a scale] — The IBS-QOL is a self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment. The IBS-QOL was measured at baseline, week 12 and week 24. The individual responses to the 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life.
  Units on a scale | 23 [4 to 62] | 20 [0 to 79] | 21.5 [0 to 79]

OUTCOME MEASURES:

1. Primary Outcome: Overall Bowel Symptom Scores (BSS)
Description: The primary end point was the overall self-reported BSS after 12 weeks of therapy for all randomized participants to assess for differences between treatment groups at the end of the treatment period (12 weeks).
  The BSS is a 100-mm visual analog scale for the different symptoms of IBS (pain/discomfort, constipation, diarrhea, and overall severity). Symptoms on the BSS can range from 0 = no pain to 100 = extreme pain.
Time Frame: After 12 weeks of treatment
Population: Analysis is based on the intention to treat (ITT) paradigm, including all randomized patients. Assuming standard deviation of the overall BSS symptom score is ~75, then 35 per group provides 80% power to detect about a 50% difference which is based on a 2-sample t-test assuming the distribution of Bowel Symptom Survey (BSS) values.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | St. John's Wort | Placebo
Number analyzed (Participants) | 35 | 35
Scores on a scale | 76 [4 to 165] | 44 [0 to 125]

2. Secondary Outcome: Bowel Symptom Score (BSS) Amongst Subgroups
Description: Median (average) BSS amongst the different IBS subgroups (diarrhea, constipation, pain, and bloating). The BSS is a 100-mm visual analog scale for the different symptoms of IBS (pain/discomfort, constipation, diarrhea, and overall severity). Symptoms on the BSS can range from 0 = no pain to 100 = extreme pain.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | St. John's Wort | Placebo
Number analyzed (Participants) | 35 | 35
Scores on a scale
  BSS for diarrhea subgroup | 32 [0 to 92] | 17 [0 to 94]
  BSS for constipation subgroup | 25.8 [0 to 78] | 16 [0 to 84]
  BSS for pain subgroup | 35.8 [1 to 77] | 23.5 [0 to 77]
  BSS for bloating subgroup | 30.3 [2 to 75] | 23.8 [1 to 70]

3. Secondary Outcome: Adequate Relief ≤ 50% During the Last 4 Weeks of Therapy
Description: Participants who reported "yes" or "no" to having adequate relief of their IBS symptoms at least 50% during the last 4 weeks of therapy.
Time Frame: Last 4 weeks of therapy
Measure: Number; unit: Percentage of Participants
Arm/Group | St. John's Wort | Placebo
Number analyzed (Participants) | 35 | 35
Percentage of Participants
  Yes | 32 | 62
  No | 50 | 26
  Missing | 18 | 12

4. Secondary Outcome: Irritable Bowel Syndrome - Quality of Life (IBS-QoL) Score
Description: The IBS-QOL is a self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment. The IBS-QOL was measured at baseline, week 12 and week 24. The individual responses to the 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life.
Time Frame: 12 weeks of treatment
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | St. John's Wort | Placebo
Number analyzed (Participants) | 35 | 35
Units on a scale | 18.8 [0.7 to 69.8] | 14.7 [1.5 to 75]

5. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D) Score
Description: We measured CES-D Score at baseline as well as bi-weekly throughout the study. The CES-D is a self-reported 20 question survey designed to measure depressive symptomatology in the general population. The possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | St. John's Wort | Placebo
Number analyzed (Participants) | 35 | 35
Units on a scale | 2 [0 to 26] | 3 [0 to 29]

6. Secondary Outcome: IBS Symptoms Moderately or a Lot Better
Description: Number of participants who stated their IBS symptoms were moderately better or a lot better at 24 weeks.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | St. John's Wort | Placebo
Number analyzed (Participants) | 35 | 35
participants
  Yes | 5 | 5
  No | 24 | 25
  Missing | 6 | 5

7. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D) Score
Description: as for outcome 5
Time Frame: 24 weeks
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | St. John's Wort | Placebo
Number analyzed (Participants) | 35 | 35
Units on a scale | 3.0 [0 to 16] | 2.5 [0 to 30]

8. Secondary Outcome: Bowel Symptom Score (BSS) at 24 Weeks
Description: The BSS is a five question, 100-mm visual analog scale of four IBS symptoms (pain/discomfort, bloating, constipation, and diarrhea), and an overall severity scale. The best possible value would be 0 (no symptoms) and the worst is 500 (severe symptoms). BSS was assessed on a bi-weekly basis.
Time Frame: 24 weeks
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | St. John's Wort | Placebo
Number analyzed (Participants) | 35 | 35
Units on a scale | 65 [12 to 149] | 60 [11 to 152]

ADVERSE EVENTS:
Time Frame: Study duration
Description: Patients will be evaluated on a bi-weekly basis by phone interview and paper questionnaire. During these queries, subjects will be asked to report study medication compliance and side effects or adverse events (AE). Adverse events will be categorized into Serious Adverse Events (SAE) and Non-serious Adverse Events (NAE).
Arm/Group | St. John's Wort | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

LIMITATIONS AND CAVEATS:
* A majority of the participants were local females with mild symptoms
* The number of participants limits power of conclusions
* We evaluated the efficacy of SJW in all subtypes of IBS not allowing specific conclusions regarding subtypes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes